CLINICAL TRIAL: NCT01756014
Title: Brain Function and Perfusion in Patients With Heart Failure
Acronym: BRAIN-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, A.A.Voors, Prof. dr., University Medical Center Groningen
Other Study IDs: BRAIN-HF
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Heart Failure; Dilated Cardiomyopathy; Perfusion; Cognitive Impairment; Cerebral Hypoperfusion
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Controls: Age matched healthy subjects
- Mild DCM: Heart failure patients with dilated cardiomyopathy (DCM) with NYHA-functional class II
- Severe DCM: Heart failure patients with dilated cardiomyopathy (DCM) with NYHA-functional class III/IV

SUMMARY:
The investigators will evaluate the determinants of cerebral impairment in patients with non-ischemic heart failure compared to controls, and its relation to cognitive function. They hypothesize that patients with heart failure have impaired brain perfusion and hemodynamic factors are associated with cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria Control Group:

* Healthy subject, as assessed by clinician
* Age matched with patient group

Exclusion Criteria Control Group:

* Age < 18 years
* Carotid artery or intracranial disease, as assessed by echo-doppler (significant stenosis > 50%)
* Unable or unwilling to undergo MRI
* The presence of ferromagnetic material in or on the body, for example tattoos with ferrous ink or pacemakers or cardiac defibrillators. Also the presence of pregnancy and claustrophobia.
* History of cognitive impairment
* Unable to understand procedures
* Unable or unwilling to provide informed consent

Inclusion Criteria DCM-group:

* Heart failure due to DCM
* 15 patients with NYHA class II
* 15 patients with NYHA class III/IV

Exclusion Criteria DCM-Group:

* Age < 18 years
* History of myocardial infarction
* History of peripheral artery disease
* History of cerebrovascular disease or
* Carotid artery or intracranial disease, as assessed by echo-doppler (significant stenosis > 50%)
* History of cognitive impairment
* Unable to undergo MRI (eg pacemaker)
* Unable to understand procedures
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients with heart failure due to dilated cardiomyopathy with NYHA II or NYHA II/IV.
  * Healthy patients
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Determinants of cerebral impairment | Baseline
  Determinants of cerebral impairment in patients with heart failure compared to controls, where cerebral impairment is defined as decreased cognitive function and cerebral hypoperfusion

SECONDARY OUTCOMES:
Prevalence of cognitive impairment | Baseline
  Prevalence of cognitive impairment in patients with heart failure
Relation of cognitive impairment with local perfusion | Baseline
  Relation of cognitive impairment with perfusion of carotid artery territory and basilar artery territory
Relation of cognitive impairment with the severity of heart failure | Baseline
  Relation of cognitive impairment with the severity of heart failure
Relation of cognitive impairment with cardiac output | Baseline
  Relation of cognitive impairment with cardiac output
Relation of cognitive impairment with the severity of congestion | Baseline
  Relation of cognitive impairment with the severity of congestion
Relation of cognitive impairment with the decrease in cerebral perfusion | Baseline
  Relation of cognitive impairment with the decrease in cerebral perfusion
The difference of cognitive domains in above relations | Baseline
  The difference of cognitive domains in above relations

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Erkelens CD, van der Wal HH, de Jong BM, Elting JW, Renken R, Gerritsen M, van Laar PJ, van Deursen VM, van der Meer P, van Veldhuisen DJ, Voors AA, Luijckx GJ. Dynamics of cerebral blood flow in patients with mild non-ischaemic heart failure. Eur J Heart Fail. 2017 Feb;19(2):261-268. doi: 10.1002/ejhf.660. Epub 2016 Nov 14. PMID 27862767